CLINICAL TRIAL: NCT01397357
Title: CARDIAC MAGNETIC RESONANCE UTILITIES IN THE EVALUATION OF ISCHEMIC HEART DISEASE: Topographical Correlation Between Ischemic Territory Injury and Coronary Angiography
Brief Title: Cardiac Magnetic Resonance Utilities in the Evaluation of Ischemic Heart Disease
Acronym: CARDIO-RM
Status: Completed | Type: Observational
Sponsor: Ettore Sansavini Health Science Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: ESREFO02
Record Dates: First submitted 2011-07-18; First posted 2011-07-19 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2015-05

CONDITIONS: Myocardial Ischemia
Keywords: Cardiac magnetic resonance; Myocardial Ischemia; Coronary Artery Disease; suspected Myocardial Ischemia
MeSH Terms: conditions — Myocardial Ischemia; Coronary Artery Disease

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- suspected Myocardial Ischemia: Patient with diagnosis of suspected coronary artery disease (CAD) or recurrent ischemic symptoms assessed by under-effort angina symptoms and/or cardiac conventional stress test, and the presence of at least two risk factors.
  Interventions: Other: Cardiac magnetic resonance - CINE MRI stress test.

INTERVENTIONS:
Other: Cardiac magnetic resonance - CINE MRI stress test. — Cardiac magnetic resonance - dipyridamole or dobutamine MRI stress test.

SUMMARY:
The purpose of this study is to evaluate CARDIAC MAGNETIC RESONANCE UTILITIES IN THE ISCHEMIC HEART DISEASE as topographical correlation between ischemic territory injury and coronary angiography.

DETAILED DESCRIPTION:
Assessing the accuracy of Cardio-RM identifying ischemic territories and their correspondence to the presence of critical coronary lesions, comparing the presence, extent and regional inducible ischaemia in the Cardiac-MRI with the presence and characteristics of vascular lesions in coronary angiography.

In particular, the study aims to evaluate the correlation between topography and function of the ischemic area revealed by the resonance and coronary artery disease documented coronary angiography.

ELIGIBILITY:
Inclusion Criteria:

1. patients with suspected ischemic heart disease or recurrent Myocardial ischemic symptoms defined as:

   * presence of:

     * chest pain related to the effort lasting 5-20 minutes, and / or
     * positive stress test for inducible Myocardial ischemia
   * presence of at least one of the following risk factors: smoke family history of cardiovascular disease hypertension dyslipidemia diabetes mellitus NID / ID
2. no contraindications to perform coronary angiography
3. informed written consent to the processing of personal and sensible data, signed and dated by the patient.

Exclusion Criteria:

* Unstable angina;
* Severe aortic stenosis
* Hypertrophic cardiomyopathy
* Pacemaker and \ or defibrillator
* Coronary stent implantation in 90 days before Cardiac MRI
* Intracranial metal clips
* Severe hypertension (systolic blood pressure> 240 mmHg, and diastolic blood pressure above 120 mmHg)
* Ventricular thrombosis and \ or atrial
* Aortic aneurysm and \ or aortic dissection
* Myocarditis, endocarditis, pericarditis
* Critical stenosis of the left notes
* State of severe anxiety or claustrophobia
* Contraindications to the use of atropine (BAV advanced glaucoma, pyloric stenosis, prostatic hypertrophy)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who refer to the clinic within 12 months, with diagnosis of suspected coronary artery disease (CAD) or recurrent ischemic symptoms assessed by under-effort angina symptoms and/or cardiac conventional stress test, and the presence of at least two risk factors.
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2011-07; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Accuracy of Cardio-RM identifying ischemic territories | 1 month
  Assessing the accuracy of Cardio-RM identifying ischemic territories and their correspondence to the presence of critical coronary lesions, comparing the presence, extent and regional inducible ischaemia in the Cardiac-MRI with the presence and characteristics of vascular lesions in coronary angiography.

SECONDARY OUTCOMES:
correlation between resonance and coronary artery disease documented coronary angiography. | 1 month
  comparison of diagnostic positivity for inducible ischemia assessed by Cardiac-MRI and the presence of coronary lesions of various degrees evaluated by coronary angiography
topographic correlation between ischemic territory and coronary lesions | 1 month
  topographic correlation between ischemic territory assessed by Cardiac-MRI and coronary lesions evaluated by coronary angiography, using the criteria defined in Sintax study and BARI study.

CONTACTS AND LOCATIONS:
Locations (1):
- Maria Cecilia Hospital, Cotignola, RA, Italy

IPD SHARING:
Plan to Share IPD: No